**STUDY TITLE:** Mind over Mood

R61 PHASE: Social Cognitive Training to Enhance the Efficacy of CBT for Depression in Youth:

A Developmental Approach

## STUDY IRB NUMBER # 190077

## PRINCIPAL INVESTIGATOR

Judy Garber, PhD., Vanderbilt University, Department of Psychology and Human Development

## **SPONSOR NAME**

National Institutes of Health (NIH) NIH Grant/Sponsor # R61 MH115125

VERSION DATE: SAP adapted from the IRB Application approved on 06/02/2019

ClinicalTrials.gov Identifier: NCT03954392

## **Statistical Analysis Plan**

We will use the general linear model (i.e., MANCOVA) to test hypotheses. The between subjects factor will be *Condition* with two levels (CBT+SCT vs. CBT only) and the within-subjects factor will be Time with two levels (baseline, post-test). We will adopt a multivariate approach to repeated measures (as assumptions of compound symmetry are untenable). Dependent variables (DVs) will vary across analyses; child age and sex, will be covariates in all analyses.

<u>Specific Aims</u>. To test whether youth in CBT+SCT have better SC skills at post-treatment than youth in CBT only at post-treatment.

Hypothesis: We will test the effect of CBT+SCT on SC skills (target) using the Faux Pau task as the DV. We will first test the 2x2 Condition x Time interaction. We expect that a 2x2 partition of this interaction will be significant, reflecting the Condition effect from baseline to post-test.

Exploratory Hypothesis: To test the effect of CBT+SCT on depressive symptoms, the DV will be the

clinician-rated depression measure (CDRS). Analyses will be the same as described for the main hypothesis except that we will test the depression measure as the dependent variable.

*Power.* To estimate power, we assumed that autocorrelations among the repeated measures were .4 - .6. With N=42 (21 per cell), alpha = .05, and a medium effect size (e.g., a .40 SD Condition effect at T2), we will have approximately .82 power to detect the initial 2x2 Condition x Time interaction ( $f_V = .32$ ). Assuming correlations of .3-.6 among the same measure over time, alpha = .05, and medium effect sizes we will have .85 power for the 2x2 Condition by Time interaction.